CLINICAL TRIAL: NCT04578106
Title: Omission of Surgery and Sentinel Lymph Node Dissection in Clinically Low-risk HER2positive Breast Cancer With High HER2 Addiction and a Complete Response Following Standard Anti-HER2-based Neoadjuvant Therapy
Brief Title: Omission of Surgery in Clinically Low-risk HER2positive Breast Cancer With High HER2 Addiction and a Complete Response Following Standard Anti-HER2-based Neoadjuvant Therapy
Acronym: ELPIS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was prematurely halted primarily due to low patient accrual. Despite efforts to optimize recruitment, the enrollment rate remained insufficient to meet the predefined targets, and continuation was deemed unfeasible
Sponsor: Fundacio Clinic Barcelona (Other)
Collaborators: SOLTI Breast Cancer Research Group (Other); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCB-ONC001 (ML41519)
Record Dates: First submitted 2020-09-29; First posted 2020-10-08 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: HER2-positive Breast Cancer; Stage I Breast Cancer
Keywords: Breast Cancer; Her2-positive; Pertuzumab; Trastuzumab; Omission surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Omission of surgery (Experimental): Neoadjuvant period: paclitaxel IV 80mg/m2 every week for 12 weeks with trastuzumab and pertuzumab Subcutaneous Fixed-Dose Combination (FDC) (a loading dose of 1200 mg pertuzumab and 600 mg trastuzumab followed by a maintenance dose of 600 mg pertuzumab and 600 mg trastuzumab once every 3 weeks) for 5 cycles. Adjuvant period: If no invasive tumor cells and no in situ disease are identified in the stereotactic-guided VAB,patients will be eligible to omit loco-regional surgery. Whole breast radiotherapy without nodal radiotherapy will then be performed. Trastuzumab and pertuzumab FDC will be continued to complete 1 year of treatment and adjuvant endocrine therapy will be indicated according to hormonal receptor status by IHC.
  Interventions: Biological: Trastuzumab and pertuzumab Subcutaneous Fixed-Dose Combination
- Surgery (No Intervention): Neoadjuvant period: paclitaxel IV 80mg/m2 every week for 12 weeks with trastuzumab and pertuzumab Subcutaneous Fixed-Dose Combination (FDC) (a loading dose of 1200 mg pertuzumab and 600 mg trastuzumab followed by a maintenance dose of 600 mg pertuzumab and 600 mg trastuzumab once every 3 weeks) for 5 cycles. Surgery: If invasive tumor cells and/or in situ disease are identified, patients will undergo surgery. Adjuvant period: All patients will continue with Trastuzumab-emtansine (T-DM1) completing 1 year of treatment (14 cycles) and adjuvant endocrine therapy will be indicated according to hormonal receptor status by IHC.

INTERVENTIONS:
Biological: Trastuzumab and pertuzumab Subcutaneous Fixed-Dose Combination — After 13 weeks of neoadjuvant treatment, a breast MRI will be performed. If a complete response is observed on breast MRI, patients will undergo a stereotactic-guided VAB of the marker area to obtain 12 cylinders of breast parenchyma, which is equivalent to 2 grams of tissue. If no invasive tumor cells and no in situ disease are identified in the stereotactic-guided VAB, patients will be eligible to omit loco-regional surgery.
  Other Names: Omission of surgery
  Arms: Omission of surgery

SUMMARY:
This is a prospective, single arm, open-label, unicenter, exploratory study in women with primary operable HER2-positive, HER2-enriched/ERBB2-high breast cancer according to PAM50 intrinsic subtype and a ERBB2 pre-defined cutoff (high vs low ERBB2 expression), to evaluate the omission of surgery and sentinel lymph node dissection in patients with HER2-E and ERBB2 high breast cancer who achieving a complete response following standard anti-HER2-based neoadjuvant therapy with paclitaxel/trastuzumab/pertuzumab. The primary trial objective is to estimate the loco-regional invasive disease-free survival at 3-year of patients who achieve a complete response based on imaging (i.e. Magnetic resonance imaging) and a stereotactic-guided vacuum-assisted breast biopsy, and omit loco-regional surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants who are at least 40 years of age on the day of signing the informed consent form with histologically confirmed diagnosis of breast cancer.
2. A participant is eligible to participate if she is not pregnant, not breastfeeding.
3. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
4. Histologically confirmed invasive adenocarcinoma of the breast, with all of the following characteristics:

   * HER2-positive status by local determination according to 2018 ASCO/CAP guidelines.
   * PAM50 HER2-enriched subtype and ERBB2-high as predefined cutoff as per central determination.
   * Unifocal invasive carcinoma: only 1 invasive focus can be observed (the tumor focus containing or not containing an in situ component)
   * Tumor largest diameter ≤4 cm as defined by breast MRI.
   * No nodal involvement (i.e. cN0). Any suspicious axillary node by ultrasound must be biopsied. If the biopsy or the FNA is negative of tumor cells, patient is eligible.
   * No evidence of distant metastasis (M0) by routine clinical assessment.
5. Patient must have known ER and PR status locally determined prior to study entry.
6. Eligible for taxane therapy.
7. Willingness of the patient to omit surgery if all criteria are met following neoadjuvant therapy.
8. Estimated life expectancy of at least 5 years irrespective of the diagnosis of breast cancer.
9. Breast cancer eligible for primary surgery
10. Have provided archival tumor tissue sample or newly obtained core. Formalin-fixed,paraffin embedded (FFPE) tissue blocks are mandatory. Available pre-treatment FFPE core biopsy evaluable for PAM50 or possibility to obtain one.
11. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
12. Ability and willingness to comply with study visits, treatment, testing and to comply with the protocol.
13. Have adequate organ function.

Exclusion Criteria:

1. Has received prior anti-cancer therapy, including investigational agents, or treatment for primary invasive breast cancer.
2. Known hypersensitivity to any of the excipients of trastuzumab, pertuzumab, TDM1 or paclitaxel.
3. Clinical stage II, III or IV.
4. History of radiotherapy in the ipsilateral breast or axilla.
5. History of surgery of the ipsilateral axilla.
6. Bilateral invasive breast cancer.
7. Infiltrating lobular carcinoma.
8. Multicentric or multifocal breast cancer, defined as the presence of two or more foci of cancer in the same or different quadrants of the same breast.
9. Patients who have undergone sentinel lymph node biopsy prior to study treatment.
10. Patient has active cardiac disease or a history of cardiac dysfunction
11. Has an active infection requiring systemic therapy.

13. Patients with a history of previous breast cancer are excluded.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aleix Prat, MD, Principal Investigator — Hospital Clinic of Barcelona; Tomas Pascual, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 20 patients were screened for the study in a single study centre (clinical setting) over the duration of 18 months. A total of 5 patients were finally selected for the study treatment after meeting all the inclusion criteria and signing the ICF
Pre-assignment Details: Out of 20 patients screened, 13 patients did not fulfill the study criteria (PAM50 subtype other than HER2-Enriched, ERBB2 high, liver metastasis, multicentric tumor).
  Finally only 5 patients that fulfilled all eligibility criteria and signed the ICF were included
Groups:
- Treatment Arm: Treatment in women with primary operable HER2-positive, HER2-enriched(HER2-E)/ERBB2-high breast cancer according to PAM50 intrinsic subtype and a ERBB2 pre-defined cutoff (high vs low ERBB2 expression):
  * Tumor size ≤ 2 cm: Paclitaxel/trastuzumab/pertuzumab (TDM-1 if residual disease)
  * Tumor size > 2 cm and ≤ 4cm: Antracycline based chemotherapy followed by Paclitaxel/trastuzumab/pertuzumab (TDM-1 if residual disease)
Period: Study treatment
Arm/Group | Treatment Arm
Started | 5
Completed | 5
Not Completed | 0
Period: Follow-up after 1 year
Arm/Group | Treatment Arm
Started | 5
Completed | 4
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: Follow up at 3 yrs
Arm/Group | Treatment Arm
Started | 4
Completed | 0
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: The baseline analysis population is the same as the treatment population
Arm/Group | Treatment Arm
Number analyzed (Participants) | 5
Age, Customized [Number; unit: participants]
  >= 40 yrs | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 5
Region of Enrollment [Number; unit: participants]
  Spain | 5
Menopausal Status [Number; unit: participants]
  Postmenopausal (min 12 mnths without menses before neoadyuvance treatment) | 4
  premenopausal | 1
ECOG baseline [Number; unit: participants] — Scale: Grades 0-4 Grade 0 - Fully active able to carry on all pre-disease performance without restriction; Grade 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature e.g. light house work office work; Grade 2 - Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours Grade 3 - Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours Grade 4 - Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  participants
    Grade 0 | 4
    Grade 1 | 1
Previous cancer history [Number; unit: participants]
  Yes | 0
  No | 5

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival at 3years
Description: To estimate the loco-regional invasive disease-free survival (LR-IDFS) at 3-year of patients who achieve a complete response based on imaging and a stereotactic-guided vacuum-assisted breast biopsy, and omit loco-regional surgery.
Time Frame: 3 years
Population: After completion of neoadjuvant therapy with paclitaxel and Trastuzumab/pertuzumab, out of 5 patients, only 3 patients showed complete response (assessed by MRI) and 2 patients (no stereo-guided VAB assessment) did not undergo surgery. However, the participants were lost to follow-up before 3-year assessments, so no evaluable 3-year survival data are available
Measure: Median (95% Confidence Interval); unit: years
Groups:
- Omision of Surgery (Complete Response): After completion of neoadjuvant therapy, if no invasive tumor cells and no in situ disease are identified in the stereotactic-guided VAB (complete response), patients will be eligible to omit loco-regional surgery
Arm/Group | Omision of Surgery (Complete Response)
Number analyzed (Participants) | 0

2. Secondary Outcome: pCR Rate
Description: rate of pathological complete response (pCR) between the treatment groups by HR status
Time Frame: pCR assessment was done following surgery after neoadjuvant therapy with paclitaxel and trastuzumzb/pertuzumab prior to adjuvant therapy
Population: While total number of HR positive patients and HR negative patients in the overall treatment group is 2 and 3 respectively, only 1 patient in the former and 2 patients in the later group were evaluated for pCR at surgery
Measure: Count of Participants; unit: Participants
Groups:
- HR Positive: patients that are hormone receptor (HR) positive (assessment at baseline)
- HR Negative: Patients that are hormone receptor (HR) negative (assessed at baseline)
Arm/Group | HR Positive | HR Negative
Number analyzed (Participants) | 1 | 2
Participants | 0 | 2

3. Secondary Outcome: Patient Reported Outcomes (Global Health Status)
Description: The EORTC QLQ-C30 was used to assess Health-Related Quality of Life (QoL). The measure consists of five functional scales (physical, role, cognitive, emotional, and social). For this study, raw scores were used without any transformation. The functional scales consist of multiple items (questions 1-28) scored on a 1-4 scale (1 = not at all, 4 = very much). Higher scores indicate worse functioning. To assess the effect of standard therapy (surgery after neoadjuvant therapy) vs. investigational therapy (omission of surgery), the global health status is reported in each of these populations before and after treatment.
  The Global Health Status (GHS) score is derived from two items (Q29 and Q30), each scored on a 1-7 scale (1 = very poor, 7 = excellent).
  Scoring method: GHS = (Q29 + Q30) / 2 Raw score range: Minimum = (1 + 1) / 2 = 1; Maximum = (7 + 7) /2 = 7
Time Frame: The questionnaire was filled by the patients at screening and post adjuvant therapy.
Population: Out of the treatment population, 3 patients underwent surgery post neoadjuvant therapy (standard therapy) and 2 patients did not undergo surgery (investigative therapy). All the patients of both the groups completed the patient reported outcomes questionaire at screening. 1 patient from the patient group that underwent surgery did not complete the questionnaire after adjuvant therapy.
Measure: Median (Full Range); unit: score on a scale
Groups:
- Patients Who Underwent Surgery (Assessment at Screening): Of the treatment population, those patients who underwent surgery post neoadjuvant therapy.
  The assessment time period is at screening
- Patients Who Underwent Surgery (Assessment After Adjuvant Therapy); Patients With Omission of Surgery (Assessment After Adjuvant Therapy): Of the treatment population, those patients who underwent surgery post neoadjuvant therapy.
  The assessment time period is after adjuvant therapy
- Patients With Omission of Surgery (Assessment at Screening): Of the treatment population, those patients with omission of surgery post neoadjuvant therapy.
  The assessment time period is at screening
Arm/Group | Patients Who Underwent Surgery (Assessment at Screening) | Patients Who Underwent Surgery (Assessment After Adjuvant Therapy) | Patients With Omission of Surgery (Assessment at Screening) | Patients With Omission of Surgery (Assessment After Adjuvant Therapy)
Number analyzed (Participants) | 3 | 2 | 2 | 2
score on a scale | 5 [5 to 6] | 4 [3.5 to 4.5] | 5.25 [4.5 to 6] | 5 [4 to 6]

ADVERSE EVENTS:
Time Frame: Study treatment duration - 1 year (neoadjuvant and adjuvant therapy)
Groups:
- Treatment Arm (Treatment With Paclitaxel); Treatment Arm (Treatment With Trastuzumab); Treatment Arm (Treatment With Pertuzumab): Treatment in women with primary operable HER2-positive, HER2-enriched(HER2-E)/ERBB2-high breast cancer according to PAM50 intrinsic subtype and a ERBB2 pre-defined cutoff (high vs low ERBB2 expression):
  * Tumor size ≤ 2 cm: Paclitaxel/trastuzumab/pertuzumab (TDM-1 if residual disease)
  * Tumor size > 2 cm and ≤ 4cm: Antracycline based chemotherapy followed by Paclitaxel/trastuzumab/pertuzumab (TDM-1 if residual disease)
- Treatment Arm (Adjuvant Treatment With TDM1): TDM-1 administered on Day 1 of a 3-week cycle q3w at a doce of 3.6 mg/kg IV as adjuvant treatment in patients of the treatment population with non-complete response in the neoadjuvant setting
Arm/Group | Treatment Arm (Treatment With Paclitaxel) | Treatment Arm (Treatment With Trastuzumab) | Treatment Arm (Treatment With Pertuzumab) | Treatment Arm (Adjuvant Treatment With TDM1)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5 | 5/5 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (Treatment With Paclitaxel) (N=5) | Treatment Arm (Treatment With Trastuzumab) (N=5) | Treatment Arm (Treatment With Pertuzumab) (N=5) | Treatment Arm (Adjuvant Treatment With TDM1) (N=3)
alopecia (Skin and subcutaneous tissue disorders) | 4 (7) | 0 (0) | 0 (0) | 0 (0)
asthenia (General disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (3)
dysguesia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 4 (4) | 0 (0)
erythema face and hands (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
erythema arms and hands (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
feet erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hands neurotoxicity (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hiporexya (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
neurotoxicity in foot (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
occasional epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
onychodystrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
onycholysis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
plantar erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
erythematous reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
muscle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
plaquetopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
decrease in hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
increase of total bilirubine (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
alat increase (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
asat increase (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
epigastralgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
increase of alkaline phosphatase (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-17): https://cdn.clinicaltrials.gov/large-docs/06/NCT04578106/Prot_SAP_000.pdf